CLINICAL TRIAL: NCT07099235
Title: Retrospective Chart Review of Patients Undergoing Intravenous Ketamine Treatments for Treatment-resistant Depression
Brief Title: Chart Review of Patients Undergoing Ketamine Treatments for Depression
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Fahad Alam, Principal Investigator, Sunnybrook Health Sciences Centre
Other Study IDs: 6828
Record Dates: First submitted 2025-07-20; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Depression - Major Depressive Disorder
Keywords: Ketamine; Major Depressive Disorder; Retrospective
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Treatment-resistant Major Depressive Disorder (MDD); DSM-5 Diagnosis of MDD
  Interventions: Drug: ketamine hydrochloride

INTERVENTIONS:
Drug: ketamine hydrochloride — Racemic ketamine is a 50/50 mixture of enantiomers (S)-ketamine and (R)-ketamine. The repeated administration of racemic ketamine intravenously at subanesthetic doses has emerged as an efficacious treatment for treatment-resistant depression.

SUMMARY:
The Ontario Ketamine and Infusion Centre (OKIC) is a CPSO-certified Level-II OHP and an outpatient centre for intravenous ketamine treatments for treatment-resistant depression. This retrospective, observational study aims to conduct a chart review on patients receiving ketamine in a naturalistic setting to develop our understanding of ketamine as an interventional approach for treatment-resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Able to provide informed consent
* Patient diagnosed with treatment-resistant depression
* Outpatient recommended and approved by psychiatrist for ketamine treatment
* Individuals who have previously received ECT, rTMS or any other neuromodulation can also receive ketamine

Exclusion Criteria:

* History of psychosis/comorbid psychiatric disorders/psychotic depression/dissociative syndromes, significant personality disorder, as clinically assessed by psychiatrist
* Using non-prescribed substance (e.g., cannabis) or alcohol use within the preceding 48 hours of treatment
* History of substance misuse and/or dependence, including chronic alcohol abuse
* Previous ketamine use
* Acute dementia/delirium
* Pregnancy/breastfeeding
* Previous sensitivity to ketamine or related compounds
* Unstable medical condition which may require anesthesia consult
* History of elevated intracranial pressure or cerebrovascular accident
* Recent (within 6 weeks) major cardiovascular event (such as myocardial infarction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with treatment-resistant depression receiving an induction phase of intravenous ketamine treatments at the OKIC from clinic opening (April 1, 2022) to June 29, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 item | Treatment Day 1 to Day 8, an average of 4 weeks.
  The PHQ-9 is a 9 item self-report assessment used to evaluate symptoms of depression. Each item has a response of 0 (None at all), 1 (Several days), 2 (More than half the days), and 3 (Nearly every day). The scale ranges from 0-27, with higher scores indicating greater severity of depression symptoms.
Beck's Depression Inventory-II | Treatment Day 1 to Day 8, an average of 4 weeks.
  The BDI-II is a 21-item self-report assessment used to evaluate symptoms of depression. Each item is scored form 0-3, with a higher score representing more severe depression. The total score ranges from 0-63, with a score >29 indicating severe depression.
Generalized Anxiety Disorder-7 item | Treatment Day 1 to Day 8, an average of 4 weeks.
  The GAD-7 is a 7 item self-report assessment used to evaluate symptoms of anxiety. Each item has a response of 0 (Not at all), 1 (Several days), 2 (More than half the days), and 3 (Nearly every day). The scale ranges from 0-21, with higher scores indicating greater severity of anxiety symptoms.

SECONDARY OUTCOMES:
Antidepressant Treatment History Form: Short Form | Baseline
  The Antidepressant Treatment History Form: Short Form (ATHF-SF) is a clinician-scored form to assess the adequacy of antidepressant treatment trials in the context of treatment-resistant depression. The form collects information regarding history of standard antidepressant medications use, such as SSRIs, SNRIs, TCAs, as well as neuromodulation and psychotherapy approaches. Previous treatments are checked off in a box, with more boxes checked meaning greater level of treatment resistance.
Adverse childhood experiences-10 item | Baseline
  The Adverse childhood experiences-10 item (ACE-10) questionnaire is a 10-item self-report assessment used to evaluate a history of adverse childhood experiences in one's life. Each item is a distinct category of an adverse childhood experience, and the 10 items are typically organized into larger categories of abuse, neglect, and family dysfunction. With a minimum score of 0 and maximum score of 10, higher scores indicate having a greater quantity of adverse childhood experiences.
Primary care PTSD screen for DSM-5 | Baseline
  The PC-PTSD-5 is a 5-item self-report assessment used to screen for probable PTSD within a primary care setting. Each item has a response option of 'Yes' or 'No.' The total score is the number of 'Yes' responses to the questions. A score of 0-3 indicates low probability of PTSD and 4 or more indicates probable PTSD.
Multidimensional Scale of Perceived Social Support scale | Baseline
  The MSPSS is a 12-item self-report assessment used to evaluate an individual's perceived level of social support. Each item has 7 response options: 1 (Very strongly disagree); 2 (Strongly disagree); 3 (Mildly disagree); 4 (Neutral); 5 (Mildly agree); 6 (Strongly agree); 7 (Very strongly agree). The score ranges from 12-84, with higher scores indicating higher levels of perceived social support.
Subject Assessment of Memory Impairment | Baseline
  The SAMI is a brief 2-part self-report assessment used to evaluate self-assessed extent of memory impairment. Part 1 asks to rate memory problems on a scale of 0-10, with 0 indicating no memory problems and 10 indicating very severe memory problems. Part 2 asks to rate the impact of these problems on their work and social activities on a scale of 1-5; 1 indicating no complaints and normal activity, and 5 indicating the symptoms to radically change their normal work and social activities.
Personal Inventory for Depression and Seasonal Affective Disorder | Baseline
  The PIDS is a 6-item self-report assessment used to evaluate seasonal affective disorder. Each item has a response of 0 (no change), 1 (slight change), 2 (moderate change), 3 (marked change), 4 (extreme change). Higher scores indicate a greater change in behaviors or feelings with the seasons.
Quick Inventory of Depressive Symptomatology-Self Report | Baseline
  The QIDS-SR is a 16-item self-report assessment used to evaluate symptoms of depression. The scoring range is from 0-27, with higher scores indicating more severe symptoms of depression.
Family history of psychiatric conditions and neurological conditions | Baseline
  Family history of health and psychiatric conditions is collected in a form with conditions alongside columns with family relationship. Individuals indicate the diagnosis of a relative for the relevant condition/ disorder by a checkmark in the appropriate box. Family history is collected for the following conditions: depression, bipolar disorder, schizophrenia, psychotic illnesses, anxiety disorder, substance abuse, suicide attempt, completed suicide, seizures, dementia, and other brain disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Ontario Ketamine and Infusion Centre - Toronto Site, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Due to patient confidentiality, individual participant data will not be shared. Only aggregate data will be published or made available.